CLINICAL TRIAL: NCT00079378
Title: A Phase I Study of Decitabine in Combination With Valproic Acid in Patients With Selected Hematologic Malignancies
Brief Title: Decitabine and Valproic Acid in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia or Previously Treated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01447; NCI-2012-01447 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6236; OSU-2003C0094; CDR0000355412; 0336 (Other: Ohio State University Medical Center); 6236 (Other: CTEP); R21CA110496 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Decitabine; Valproic Acid

ARMS (1):
- Treatment (decitabine, valproic acid) (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 or 1-10. Treatment repeats every 28 days.
  Cohorts of 6 patients receive escalating doses of decitabine until the MEPD is determined. The MEPD is defined as the dose at which at least 5 of 6 patients meet gene methylation criteria and no more than 1 of 6 patients experiences DLT.
  Once the MEPD is determined, patients receive decitabine at that dose level administered as above and oral valproic acid three times daily on days 5-21. Treatment repeats every 28 days.
  Cohorts of 3-6 patients receive escalating doses of valproic acid until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. The MEPD of valproic acid is then determined using established gene methylation and toxicity criteria. Treatment continues for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: decitabine; Drug: valproic acid; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Drug: valproic acid — Given orally
  Other Names: Alti-Valproic; Depakene; Novo-Valproic; VA
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine and valproic acid in treating patients with refractory or relapsed acute myeloid leukemia or previously treated chronic lymphocytic leukemia or small lymphocytic leukemia. Drugs used in chemotherapy, such as decitabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Valproic acid may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Combining decitabine with valproic acid may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the minimally effective pharmacological dose (MEPD) of decitabine in patients with refractory or relapsed acute myeloid leukemia or with previously treated chronic lymphocytic lymphoma or small lymphocytic lymphoma.

II. Determine the maximum tolerated dose (MTD) of valproic acid in combination with the MEPD of decitabine in these patients.

III. Determine the MEPD of valproic acid in combination with decitabine in these patients.

IV. Determine the qualitative and quantitative toxic effects of decitabine alone and in combination with valproic acid, in terms of organ specificity, time course, predictability, and reversibility in these patients.

SECONDARY OBJECTIVES:

I. Determine the therapeutic response in patients treated with decitabine alone and in combination with valproic acid.

II. Determine the pharmacokinetics of this regimen in these patients. III. Determine kinetics of methyltransferase activity and re-expression of select target genes in AML [p15, estrogen receptor (ER), WT-1, calcitonin, MYOD1] and in CLL/SLL [DERMO-1, DAPK, and ID4] known to be methylated in primary tumor cells.

IV. Correlate baseline and post-treatment changes in DNA methyltransferases (MT1, MT3a, and MT3b) expression with achievement of decitabine MEPD, toxicity, treatment resistance, and disease response in these patients.

V. Determine kinetics of HDAC enzyme inhibition and changes in the acetylation status of histones H3 or H4 following treatment with the combination. These parameters will be used to define the MEPD of the combination.

VI. Examine baseline and post-therapy changes in the "histone code' in both AML and CLL cells by assessment of the acetylation and methylation status of histones H3 and H4 lysine residues using both Western Blot and Mass Spectrometry techniques.

OUTLINE: This is a dose-escalation study. Patients are stratified according to disease (refractory or relapsed acute myeloid leukemia vs chronic lymphocytic leukemia or small lymphocytic lymphoma).

Patients receive decitabine IV over 1 hour on days 1-5 or 1-10. Treatment repeats every 28 days.

Cohorts of 6 patients receive escalating doses of decitabine until the minimally effective pharmacological dose (MEPD) is determined. The MEPD is defined as the dose at which at least 5 of 6 patients meet gene methylation criteria and no more than 1 of 6 patients experiences dose-limiting toxicity (DLT).

Once the MEPD is determined, patients receive decitabine at that dose level administered as above and oral valproic acid three times daily on days 5-21. Treatment repeats every 28 days.

Cohorts of 3-6 patients receive escalating doses of valproic acid until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. The MEPD of valproic acid is then determined using established gene methylation and toxicity criteria. Treatment continues for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML (Stratum I) or CLL/SLL (Stratum II) will be enrolled
* Patients in stratum I will have one of the following:

  * Primary refractory or relapsed (in 1 year or less) disease and not a candidate for potentially curative therapy
  * Untreated AML patients who are not candidates for chemotherapy
  * Patients in stratum I must have a normal WBC (=< 10 x 10^9/L) or a WBC =< 40 x 10^9/L that is stable for 1 week (this may be sustained with hydroxyurea prior to starting therapy and during the first 4 days of therapy if clinically indicated)
* Patients in stratum II will have received at least one prior therapy for CLL/SLL that has included a purine analog; patients in stratum II with a history of severe autoimmune disease or requiring therapy with chronic corticosteroids or who have any other specific relative contraindications to receive a purine analog and, therefore, have received another form of therapy that include alkylating agents will be eligible to participate
* Performance status - ECOG 0-2
* At least 12 weeks life expectancy
* Stratum II:

  * No uncontrolled autoimmune hemolytic anemia
  * No idiopathic thrombocytopenia purpura
* Bilirubin =< 1.5 mg/dL
* ALT and AST =< 2 times upper limit of normal
* Creatinine =< 2.0 mg/dL
* No active infection requiring IV antibiotics
* HIV negative
* No other severe medical condition that would preclude study participation
* No psychiatric condition that would preclude study compliance
* No history of seizures
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 14 days since prior chemotherapy (except hydroxyurea)
* No prior FR901228 (depsipeptide) for step 2 of this study
* No other concurrent chemotherapy
* No concurrent corticosteroids for antiemetic therapy
* No concurrent hormonal therapy except for the following:

  * Steroids for treatment of adrenal failure or septic shock
  * Insulin for diabetes
  * Tamoxifen or equivalent for breast cancer prevention or adjuvant therapy
  * Estrogens or progestins for gynecologic indications
* More than 14 days since prior radiotherapy
* No concurrent palliative radiotherapy
* No concurrent anticonvulsant medication, including valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-02; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
MEPD of single agent decitabine | 10 days
MTD of the combination of valproic acid with the MEPD of decitabine | Up to 21 days
MEPD of valproic acid in combination with decitabine | Up to 29 days
Qualitative and quantitative toxicities of single agent decitabine alone and in combination with valproic acid in regard to organ specificity, time course, predictability, and reversibility | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Blum W, Klisovic RB, Hackanson B, Liu Z, Liu S, Devine H, Vukosavljevic T, Huynh L, Lozanski G, Kefauver C, Plass C, Devine SM, Heerema NA, Murgo A, Chan KK, Grever MR, Byrd JC, Marcucci G. Phase I study of decitabine alone or in combination with valproic acid in acute myeloid leukemia. J Clin Oncol. 2007 Sep 1;25(25):3884-91. doi: 10.1200/JCO.2006.09.4169. Epub 2007 Aug 6. PMID 17679729